CLINICAL TRIAL: NCT02184416
Title: AXITINIB IN ADVANCED / METASTATIC RENAL CELL CARCINOMA - A NON-INTERVENTIONAL STUDY OF REAL WORLD TREATMENT OUTCOMES IN PATIENTS RECEIVING 2ND LINE AXITINIB AFTER 1ST LINE SUNITINIB (ADONIS)
Brief Title: Study Of The Impact Of Inlyta In 2nd Line On The Treatment Outcomes Of mRCC Patients Treated With Sutent In 1st Line In The Real Life Setting
Acronym: ADONIS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061078; ADONIS (Other: Alias Study Number)
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Renal Cell Carcinoma (mRCC)
Keywords: Inlyta; axitinib; Sutent; sunitinib; renal
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Watchful Waiting; Sorafenib; pazopanib; Everolimus; temsirolimus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Arm: Patients will be enrolled when they start a treatment with Sutent in 1st line or Inlyta in 2nd line post Sutent treatment. The possible sequences of treatment under investigation will be:
  * Sutent (prospective) - Inlyta
  * Sutent (retrospective) - Inlyta
  * Sutent - not further active treatment (supportive care)
  * Sutent - other second line treatment (Nexavar (sorafenib), Votrient (pazopanib), Afinitor (everolimus), Torisel (temsirolimus), other))
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — The study is non interventional. All drugs will be prescribed
  Other Names: Nexavar (sorafenib), Votrient (pazopanib), Afinitor (everolimus), Torisel (temsirolimus)

SUMMARY:
This is an international, multi-centre, prospective (partly retrospective), observational study to evaluate treatment patterns and clinical outcomes in patients with advanced or metastatic RCC treated with sunitinib in first line and/or receiving axitinib in second line post sunitinib. The study is designed to enroll approximately 750 patients over the course of an enrollment period of approximately 36 months.

DETAILED DESCRIPTION:
Patients will be enrolled when they start a treatment with Sutent in 1st line or Inlyta in 2nd line post Sutent treatment. The possible sequences of treatment under investigation will be:

* Sutent (prospective) - Inlyta
* Sutent (retrospective) - Inlyta
* Sutent - not further active treatment (supportive care)
* Sutent - other second line treatment (Nexavar (sorafenib), Votrient (pazopanib), Afinitor (everolimus), Torisel (temsirolimus), other)) The study will enroll approximately 750 adv/mRCC patients at the 1st and 2nd line treatment level. Patients will be enrolled when they start a treatment with Sutent in 1st line or Inlyta in 2nd line post Sutent treatment. Therefore for some patients there will be a retrospective Sutent data collection. The primary endpoints of this study in patients with adv/mRCC are PFS and TTF for patients receiving Inlyta in 2nd line, and the combined PFS and TTF for patients receiving the Sutent-Inlyta sequence. In this non-interventional real life study, the objective is only descriptive and the sample size will rely on the precision of the estimate.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age and over
* Histologically confirmed diagnosis of advanced/metastatic renal carcinoma (clear cell RCC as well as non-clear cell RCC) with measurable disease according to RECIST 1.1
* Patients being treated with Sutent in 1st line according to the European therapeutic indication and/or being treated with Inlyta in 2nd line according to the European approved therapeutic indication (except post cytokines)
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients being treated with cytokines or any other treatment outside of Sutent in 1st line
* Patients receiving anti -tumor treatment beyond a second line
* Patients already under Sutent, already under Inlyta: enrolment must occur at the beginning of each line of treatment (before or at the first follow up visit at the latest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll adv/mRCC patients when they start a treatment with Sutent in 1st line or Inlyta in 2nd line post Sutent treatment.
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 60 months
  PFS for patients with adv/mRCC receiving Inlyta in 2nd line post Sutent is defined as the time from when the patient receives the first dose of Inlyta to the time of progression or death due to any cause, whichever occurs first
Progression-Free Survival (PFS) | 60 months
  Combined PFS for patients with adv/mRCC receiving the Sutent-Inlyta sequence is defined as the time from when the patient receives the first dose with Sutent in first line, until progression or death due to any cause with Inlyta in 2nd line, whichever occurs first during the Sutent-Inlyta sequence
Time to Treatment Failure (TTF) | 60 months
  TTF for Inlyta 2nd line is defined as from when the patient receives the first dose of Inlyta to the time of Inlyta discontinuation (date completed by the physician).
Time to Treatment Failure (TTF) | 60 months
  TTF for the Sutent-Inlyta sequence is defined as the time from when the patient receives the first dose with Sutent in first line to the time of Inlyta discontinuation (date completed by the physician).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 60 months
  ORR for adv/mRCC patients receiving Inlyta in 2nd line post Sutent defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR) according to RECIST criteria v1.1, relative to all patients who have baseline measurable disease.
Overall Survival (OS) | 60 months
  OS for adv/mRCC patients receiving Sutent in first line followed by Inlyta in 2nd line as measured from the date of first Sutent dose to the date of death of any cause.
Time to strategy failure (TSF) | 60 months
  TSF for patients receiving the Sutent-Inlyta sequence is defined as the time from when the patient receives the first dose with Sutent in first line to the time of Inlyta discontinuation (date completed by the physician) without the time between discontinuation of Sutent and start of Inlyta.
Dosing | 60 months
  Description of real life usage of flexible dosing across Europe with description of treatment schedules (dosing change, dosing schedule, average dose received during the period treatment)
Proportion of titrated patients | 60 months
  A patient is considered as titrated when an Inlyta dose increase is maintained for at least 4 weeks.
Progression-Free Survival (PFS) | 60 months
  PFS for titrated and non-titrated patients when they receive Inlyta in 2nd line post Sutent
Efficacy | 60 months
  Efficacy parameters (PFS, OS) for the combined 1st line Sutent - 2nd line sequences according to the second line post Sutent (other than Sutent-Inlyta)
Safety | 60 months
  Safety description with AE listing in patients receiving Inlyta
QoL | 60 months
  QoL using the Functional Assessment of Cancer Therapy-Kidney Symptom Index 19 (FKSI-19) questionnaire and the Mental Health (MH) and Role-Emotional (RE) domains of the SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (110):
- Austria (8):
  - Landeskrankenhaus Bregenz, Bregenz
  - AKh Linz, Linz
  - Krankenhaus der Barmherzigen Schwestern Linz Abteilung fuer Urologie, Linz
  - Krankenhaus Oberwart, Oberwart
  - Universitasklinik für Urologie und Andrologie, Salzburg
  - AKH - Universitaetsklinik fuer Innere Medizin I, Vienna
  - AKH-Universitat Klinik fur Innere Medizin I, Vienna
  - Sozialmedizinisches Zentrum Ost, Vienna
- Belgium (5):
  - ASZ Aalst - Campus Aalst, Aalst
  - Imeldaziekenhuis, Bonheiden
  - Algemeen Ziekenhuis Sint-Lucas, Dienst Oncologie, Ghent
  - AZ Maria Middelares, Ghent
  - Clinique St Pierre - Oncologie, Ottignies
- France (57):
  - Centre Antoine Lacassagne, Service d'Oncologie, Nice, Alpes-maritimes
  - Cl du Docteur Calabet / Cromg, Agen
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Department Oncologie, Medecine Interene, Avignon
  - Centre d'Oncologie et de Radiotherapie du pays Basque, Bayonne
  - Clinique Bordeaux Tivoli Ducos, Bordeaux
  - Hôpital Saint-André, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier De Bourg En Bresse - Hopital Fleyriat, Bourg-en-Bresse
  - Centre Catalan Urologie Andrologie, Cabestany
  - C.H.G. Antoine Gayraud, Medecine Interne, Carcassonne
  - CH Rene Dubos, Cergy-Pontoise
  - Hopital Prive Sainte Marie, Chalon-sur-Saône
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Pole Sante Republique, Clermont-Ferrand
  - Centre d'Oncologie du Parc, Dijon
  - Clinique Clement Drevon, Dijon
  - Clinique Sainte Marguerite, Hyères
  - Hopital prive La Louviere, Lille
  - Hopital Dupuytren - Oncologie Medicale, Limoges
  - Centre Hospitalier de Longjumeau, Longjumeau
  - Clinique de la Sauvegarde, Lyon
  - Centre Hospitalier Prive Clairval, Marseille
  - Hopital Timone Adultes, Marseille
  - Hopital Nord, Marseille
  - Hopital Belle-Isle, Metz
  - Hopital Clinique Claude-Bernard, Metz
  - Groupe Hospitalier Intercommunal le Raincy Montfermeil, Montfermeil
  - Clinique Clémentville - Oncologie, Montpellier
  - Centre d'Oncologie de Gentilly, Nancy
  - Centre d'Oncology de Gentilly, Nancy
  - Hôpital Universitaire Carémeau, Nîmes
  - Centre Hospitalier de Pau, Pau
  - Polyclinique de Francheville, Périgueux
  - Centre Hospitalier Lyon Sud - Service d oncologie medicale, Pierre-Bénite
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CH Annecy Genevois, Pringy
  - CHR Annecy, Pringy
  - Institut Jean Godinot, Reims
  - Cl Armoricaine Radiologie / Radiotherapie, Saint-Brieuc
  - CHP Saint Gregoire, Saint-Grégoire
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
  - Centre Rene Gauducheau - Service Oncologie Medicale, Saint-Herblain
  - Pôle Hospitalier Mutualiste, Saint-Nazaire
  - Groupe Hospitaier Sud Reunion, Saint-Pierre
  - Centre Hospitalier Sud Reunion, Saint-Pierre-des-Corps
  - Centre de Radiothérapie,, Strasbourg
  - Hopital de Hautepierre-Service Oncologie at Hematologie, Strasbourg
  - Hopital FOCH, Suresnes
  - Hopital Georges Pianta, Thonon-les-Bains
  - Hopital Sainte Musse, Toulon
  - Centre Hospitalier du Marechal Juin, Valence
  - Clinique les Dentellieres, Valenciennes
  - Hopital Jean BERNARD - Tours - 7eme etage, Valenciennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- General Hospital of Chest Diseases of Athens "Sotiria", Athens, Greece
- Italy (6):
  - IRCC Oncologia Medica, Candiolo (TO)
  - Divisione di Oncologia Medica, Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola (FC)
  - Istituto Nazionale Tumori, Oncologia Medica B, Milan
  - Divisione di Oncologia, AORN Antonio Cardarelli, Napoli
  - Istituto per lo Studio e la Cura dei Tumori Fondazione Pascale, Napoli
  - IRCCS Policlinico San Matteo, Pavia
- Viecuri Medical Centre, BL Venlo, Netherlands
- Spain (24):
  - Consorcio Hospitalario Parc Tauli, Sabadell, Barcelona
  - Hospital de Navarra, Pamplona, Navarre
  - Complexo Hospitalario Universitario A Coruña. Hospital Teresa Herrera, A Coruña
  - Hospital Principe de Asturias, Alcalá de Henares
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Sant Pau, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Yague, Burgos
  - Institut Catala Oncologia - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital de Leon, León
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Servicio de Oncologia Medica, Madrid
  - Hospital Morales Meseguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Virgen de La Salud, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia
  - Salud Hospital Universitario Dr. Peset, Valencia
  - Centro Sanitario Hospital Universitario y Politecnico La Fe, Valencia
  - Centro Médico, Vigo
  - H. U. de Vigo- Hospital Álvaro Cunqueiro/Servicio de Oncologia Medica, Vigo
- United Kingdom (8):
  - Consultant Oncologist, Cheltenham, Gloustershire
  - Kent & Canterbury Hospital, Canterbury, KENT
  - Royal Surrey County Hospital, Guildford, Surrey
  - Department of Cancer Medicine, Dundee, Tayside
  - Royal United Hospital Bath NHS, Bath
  - Department of Academic Oncology, Cottingham
  - Royal Marsden Hospital, Royal Marsden NHS Foundation Trust, London
  - Christie Hospital NHS Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061078&StudyName=Study%20Of%20The%20Impact%20Of%20Inlyta%20In%202nd%20Line%20On%20The%20Treatment%20Outcomes%20Of%20mRCC%20Patients%20Treated%20With%20Sutent%20In%201st%20Line%20In%20The%20Re

DOCUMENTS (2):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02184416/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02184416/SAP_001.pdf